CLINICAL TRIAL: NCT00083070
Title: A Phase I Trial Of Temozolomide In Pediatric Patients With Refractory/Recurrent Leukemias
Brief Title: Temozolomide in Treating Young Patients With Refractory or Recurrent Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL0411; CDR0000362059 (Other: Clinical Trials.gov); COG-ADVL0411 (Other: Children's Oncology Group)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; relapsing chronic myelogenous leukemia; childhood acute promyelocytic leukemia (M3); blastic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide Therapy (Experimental)
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide
  Other Names: Temodar; NSC # 362856

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of temozolomide in treating young patients with refractory or recurrent leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of temozolomide in pediatric patients with refractory or recurrent leukemia.
* Determine the toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

Secondary

* Determine the antitumor activity of this drug in these patients.
* Determine the biologic activity and mechanism(s) of resistance to this drug in these patients.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3-36 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed leukemia of any of the following types:

  * Acute lymphoblastic leukemia
  * Acute myeloid leukemia
  * Chronic myelogenous leukemia in blast crisis
* Refractory or recurrent disease
* Immunophenotypic confirmation of disease at initial diagnosis or recurrence
* More than 25% blasts in the bone marrow (M3)
* Active extramedullary disease allowed except for leptomeningeal disease
* No known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* No active CNS disease

PATIENT CHARACTERISTICS:

Age

* 1 to 21

Performance status

* Karnofsky 50-100% (for patients > 10 years of age)
* Lansky 50-100% (for patients ≤ 10 years of age)

Life expectancy

* Not specified

Hematopoietic

* WBC < 30,000/mm^3 (hydroxyurea or leukapheresis allowed at the discretion of the principal investigator)
* Platelet count ≥ 20,000/mm^3 (platelet transfusions allowed)
* Hemoglobin ≥ 8.0 g/dL (red blood cell transfusions allowed)

Hepatic

* ALT ≤ 5 times upper limit of normal (ULN)
* Albumin ≥ 2 g/dL
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine normal for age OR
* Creatinine clearance OR radioisotope glomerular filtration rate ≥ 70 mL/min/1.73 m^2

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 7 days since prior biologic therapy, including immunotherapy
* At least 3 months since prior stem cell transplantation

  * No evidence of active graft-vs-host disease
* No concurrent biologic therapy
* No concurrent immunotherapy

Chemotherapy

* Recovered from prior chemotherapy
* At least 6 weeks since prior nitrosoureas
* Prior therapy with hydroxyurea allowed for up to 24 hours before initiation of study drug
* No other concurrent chemotherapy

Endocrine therapy

* Concurrent hydrocortisone or other corticosteroids allowed as premedications prior to blood product transfusions in patients with prior severe allergic reactions

Radiotherapy

* Recovered from prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No other concurrent anticancer agents
* No other concurrent investigational drugs

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2004-03; Primary Completion 2004-09 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose
Toxicity as assessed by CTCAE 3.0
Pharmacokinetics as assessed by CI, area under the curve (AUC), and half-life (T ½)

SECONDARY OUTCOMES:
Antitumor activity
Biologic activity and mechanisms of resistance

CONTACTS AND LOCATIONS:
Overall Officials: Terzah M. Horton, MD, PhD, Study Chair — Texas Children's Cancer Center
Locations (16):
- United States (14):
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Horton TM, Thompson PA, Berg SL, Adamson PC, Ingle AM, Dolan ME, Delaney SM, Hedge M, Weiss HL, Wu MF, Blaney SM; Children's Oncology Group Study. Phase I pharmacokinetic and pharmacodynamic study of temozolomide in pediatric patients with refractory or recurrent leukemia: a Children's Oncology Group Study. J Clin Oncol. 2007 Nov 1;25(31):4922-8. doi: 10.1200/JCO.2007.12.0667. PMID 17971589
- [Result] Horton TM, Dolan E, Hegde M, et al.: A phase I study of temozolomide (Temodar®) in pediatric patients with relapsed or refractory leukemia: a Children's Oncology Group study. [Abstract] Blood 106 (11): A-4455, 2005.